CLINICAL TRIAL: NCT06405165
Title: The Effect of Flipped-Jigsaw Learning Models on Learning Knowledge and Skills for Urinary Catheter Care in Nursing Students
Brief Title: Jigsaw Learning Model and Urinary Catheter Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Aysun Acun 7
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-06

CONDITIONS: The Effect of the Flipped-Jigsaw Learning Model on Learning
Keywords: flipped training; Jigsaw learning model; nursing students; urinary catheter care

STUDY DESIGN:
Intervention Model Description: The effect of the flipped education-Jigsaw learning model on the knowledge level of urinary catheter care in nursing students.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Knowledge level of nursing students (Experimental)
  Interventions: Other: student success
- Effect of flipped education-Jigsaw learning model (Experimental)
  Interventions: Other: student success

INTERVENTIONS:
Other: student success — The effect of the flipped education-Jigsaw learning model on the knowledge level of urinary catheter care in nursing students.

SUMMARY:
This study was planned to evaluate the effect of the reversed Jigsaw learning model on urinary catheter care in nursing students. It is anticipated that the relevant method will increase the knowledge level of students.

DETAILED DESCRIPTION:
In this research, it is aimed to use the flipped learning model and the Jigsaw learning model together. The group in which the intervention will be carried out will continue their education outside the classroom with videos and lecture notes, and will carry out group work during class time as required by the Jigsaw strategy. In a study in which these two teaching methods were applied to nursing students within the scope of an ethics course, an increase in the students; ethical sensitivity and familiarity with ethical dilemmas was noted. Therefore, in this study focusing on urinary catheter care, the academic success of the students will make a difference in patient safety. It is anticipated that this study is original in its field and will guide instructors within the scope of teaching techniques.

ELIGIBILITY:
Inclusion Criteria:

* Getting information about urinary catheter care for the first time
* Volunteering to participate in the study

Exclusion Criteria:

* Having received previous training on urinary catheter care
* Not volunteering to participate in the study
* Not participating in the posttest and follow-up test

Ages: 17 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
The effect of the flipped education-Jigsaw learning model on the knowledge level of urinary catheter care in nursing students. | 5 weeks for each participant

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Bilecik, Turkey (Türkiye)